CLINICAL TRIAL: NCT05886777
Title: A STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF COMBINED VACCINE CANDIDATE(S) AGAINST INFECTIOUS RESPIRATORY ILLNESSES, INCLUDING COVID-19 AND RSV, IN HEALTHY INDIVIDUALS
Brief Title: A Study to Learn About Two or More Vaccines That Are Put Together as One Shot Against Infectious Lung Illnesses, Including COVID-19 and Respiratory Syncytial Virus (RSV).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C5481001
Record Dates: First submitted 2023-05-31; First posted 2023-06-02 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: SARS-CoV-2; COVID-19; Flu; Influenza; Vaccine; RSV; Respiratory Syncytial Virus; Combination vaccine; mRNA vaccine
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1 (Experimental): Combination [RSVpreF+BNT162b2] + Quadrivalent influenza vaccine (QIV)
  Interventions: Biological: Combination [RSVpreF+BNTb162b2]; Biological: QIV
- Group 2 (Experimental): Combination [RSVpreF+BNT162b2] + placebo
  Interventions: Biological: Combination [RSVpreF+BNTb162b2]; Biological: Normal Saline Placebo
- Group 3 (Active Comparator): BNT162b2 + placebo
  Interventions: Biological: Bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: Normal Saline Placebo
- Group 4 (Active Comparator): RSVpreF + placebo
  Interventions: Biological: RSVpreF; Biological: Normal Saline Placebo
- Group 5 (Active Comparator): QIV + placebo
  Interventions: Biological: QIV; Biological: Normal Saline Placebo
- Group 6 (Experimental): Coadministration RSVpreF + bivalent BNT162b2 + placebo
  Interventions: Biological: Bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: RSVpreF; Biological: Normal Saline Placebo
- Group 7 (Experimental): Coadministration RSVpreF + bivalent BNT162b2 + QIV
  Interventions: Biological: Bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: RSVpreF; Biological: QIV

INTERVENTIONS:
Biological: Combination [RSVpreF+BNTb162b2] — Combination of RSVpreF and Bivalent BNT162b2 given as a single intramuscular injection
  Arms: Group 1; Group 2
Biological: Bivalent BNT162b2 (original/Omi BA.4/BA.5) — Bivalent BNT162b2 given as an intramuscular injection
  Arms: Group 3; Group 6; Group 7
Biological: RSVpreF — RSVpreF given as an intramuscular injection
  Arms: Group 4; Group 6; Group 7
Biological: QIV — Licensed QIV given as an intramuscular injection
  Arms: Group 1; Group 5; Group 7
Biological: Normal Saline Placebo — Normal saline (0.9% sodium chloride solution for injection)
  Arms: Group 2; Group 3; Group 4; Group 5; Group 6

SUMMARY:
The purpose of the study is to learn about the safety and effects of a combined vaccine for RSV and COVID-19 when given with a seasonal flu vaccine or when given alone. A combined vaccine will help to reduce the number of vaccinations given when trying to prevent respiratory infections.

This study is seeking participants who:

* are 65 years of age or older.
* are healthy or have well-controlled chronic conditions.
* in the past have received at least 3 US-authorized mRNA COVID 19 vaccines, with the most recent vaccine being an updated booster vaccine given at least more than or equal to 150 days before Visit A101 (Day 1).
* have not had a flu shot in the last 120 days.
* agree to be present for all study visits, procedures, and blood draws.

Participants will be involved in this study for 6 months. During this time, participants will have 2 study visits at the study clinic and a 6-month telephone contact.

ELIGIBILITY:
Substudy A Inclusion Criteria:

1. Male or female participants ≥65 years of age at Visit 1 (Day 1).
2. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
4. Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
5. Participants who have received at least 3 prior US authorized mRNA COVID 19 vaccines, with the last dose being an updated (bivalent) vaccine given at least ≥150 days before Visit A101 (Day 1).

Substudy A Exclusion Criteria:

1. A confirmed diagnosis of COVID 19, RSV infection, or influenza ≤120 days before study intervention administration.
2. History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
3. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
4. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
5. Allergy to egg proteins (egg or egg products) or chicken proteins.
6. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
7. Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before enrollment through conclusion of the study.
8. Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or planned receipt throughout the study.
9. Receipt of any RSV vaccine at any time prior to enrollment, or planned receipt throughout the study.
10. Receipt of any influenza vaccine ≤120 days before study enrollment.
11. Participation in other studies involving a study intervention within 28 days before randomization. Anticipated participation in other studies within 28 days after receipt of study intervention in this study.
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1142 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (37):
  - West Coast Research, Dublin, California
  - Marvel Clinical Research, Huntington Beach, California
  - Orange County Research Center, Lake Forest, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Research Foundation, San Diego, California
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Wr-Msra.Llc, Lake City, Florida
  - Optimal Research, Melbourne, Florida
  - Suncoast Research Group, Miami, Florida
  - Clinical Site Partners, LLC dba CSP Orlando, Winter Park, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Great Lakes Clinical Trials - Gurnee, Gurnee, Illinois
  - Optimal Research, Peoria, Illinois
  - Bio-Kinetic Clinical Applications LLC DBA QPS_MO (Patient Screening Only), Springfield, Missouri
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications, LLD dba QPS-MO, Springfield, Missouri
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Headlands Horizons LLC, Brownsville, Texas
  - DM Clinical Research - Cy Fair, Houston, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - DM Clinical Research, Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Virginia Research Center, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Neutel JM, Erdem R, Jiang Q, Cannon K, Stacey H, Newton R, Gomme E, Li W, Mensa FJ, Tureci O, Sahin U, Swanson KA, Munjal I, Cooper D, Koury K, Anderson AS, Gurtman A, Kitchin N; C5481001 Study Group. Safety and Immunogenicity of Concomitant Administration and Combined Administration of Bivalent BNT162b2 COVID-19 Vaccine and Bivalent RSVpreF Respiratory Syncytial Virus Vaccine with or Without Quadrivalent Influenza Vaccine in Adults >/= 65 Years of Age. Vaccines (Basel). 2025 Feb 5;13(2):158. doi: 10.3390/vaccines13020158. PMID 40006705
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5481001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1142 participants were enrolled in this study, 1083 participants were randomized to receive study vaccination, out of which, 1073 participants were vaccinated.
Pre-assignment Details: Participants were randomized to receive combined respiratory syncytial virus stabilized prefusion F subunit vaccine (RSVpreF) and bivalent BNT162b2 (original/Omi BA.4/BA.5) vaccine [RSVpreF + BNT162b2], administered concomitantly with a seasonal quadrivalent influenza vaccine (QIV) or placebo.
Groups:
- Group 1: [RSVpreF + BNT162b2] + QIV: Participants were randomized to receive combination of RSVpreF and Bivalent BNT162b2 as a single intramuscular injection along with concomitant QIV as intramuscular injection on Day 1.
- Group 2: [RSVpreF+BNT162b2] + Placebo: Participants were randomized to receive combination of RSVpreF and Bivalent BNT162b2 as a single intramuscular injection along with placebo as intramuscular injection on Day 1.
- Group 3: BNT162b2 + Placebo: Participants were randomized to receive BNT162b2 as a single intramuscular injection along with placebo as intramuscular injection on Day 1.
- Group 4: RSVpreF + Placebo: Participants were randomized to receive RSVpreF as a single intramuscular injection along with placebo as intramuscular injection on Day 1.
- Group 5: QIV + Placebo: Participants were randomized to receive QIV as a single intramuscular injection along with placebo as intramuscular injection on Day 1.
- Group 6: RSVpreF + BNT162b2 + Placebo: Participants were randomized to receive RSVpreF + BNT162b2 + Placebo as a single intramuscular injection on Day 1.
- Group 7: RSVpreF + BNT162b2 + QIV: Participants were randomized to receive RSVpreF + BNT162b2 + QIV as a single intramuscular injection on Day 1.
Period: Overall Study
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV
Started | 155 | 154 | 152 | 155 | 151 | 158 | 158
Completed | 153 | 151 | 147 | 150 | 148 | 155 | 157
Not Completed | 2 | 3 | 5 | 5 | 3 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1 | 0 | 2 | 0
Not completed — Other | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 4 | 3 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV | Total
Number analyzed (Participants) | 155 | 154 | 152 | 155 | 151 | 158 | 158 | 1083
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (5.36) | 71.7 (5.01) | 71.1 (4.70) | 72.1 (4.69) | 72.3 (5.12) | 71.3 (4.87) | 71.6 (4.79) | 71.7 (4.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 94 | 81 | 81 | 81 | 95 | 83 | 603
  Male | 67 | 60 | 71 | 74 | 70 | 63 | 75 | 480
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 15 | 11 | 18 | 12 | 18 | 15 | 110
  Not Hispanic or Latino | 134 | 138 | 140 | 137 | 139 | 139 | 142 | 969
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 4
  Asian | 8 | 4 | 2 | 1 | 3 | 3 | 5 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 10 | 12 | 13 | 10 | 9 | 14 | 13 | 81
  White | 135 | 138 | 133 | 143 | 136 | 140 | 138 | 963
  More than one race | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions included pain, redness and swelling at the injection site, recorded by participants in an electronic diary (e-diary). Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity and severe: prevented daily activity. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 centimeter (cm) and graded as mild: 2.5 cm to 5.0 cm; moderate: greater than (>) 5.0 cm to 10.0 cm; severe: > 10 cm.
Time Frame: Day 1 to Day 7 after Vaccination on Day 1
Population: Safety population included all participants who received the study intervention. Here, "Number of Participants Analyzed" signifies number of participants reporting at least 1 response in the e-diary.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV
Number analyzed (Participants) | 154 | 153 | 150 | 152 | 149 | 157 | 158
Percentage of participants
  Pain at the injection site: Mild | 49.4 [41.2 to 57.5] | 45.8 [37.7 to 54.0] | 54.7 [46.3 to 62.8] | 10.5 [6.1 to 16.5] | 48.3 [40.1 to 56.6] | 45.2 [37.3 to 53.4] | 44.9 [37.0 to 53.0]
  Pain at the injection site: Moderate | 7.8 [4.1 to 13.2] | 5.9 [2.7 to 10.9] | 7.3 [3.7 to 12.7] | 0 [0.0 to 2.4] | 3.4 [1.1 to 7.7] | 11.5 [6.9 to 17.5] | 7.6 [4.0 to 12.9]
  Pain at the injection site: Severe | 0 [0.0 to 2.4] | 0.7 [0.0 to 3.6] | 0.7 [0.0 to 3.7] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.3] | 1.3 [0.2 to 4.5]
  Redness: Mild | 3.2 [1.1 to 7.4] | 5.9 [2.7 to 10.9] | 5.3 [2.3 to 10.2] | 1.3 [0.2 to 4.7] | 2.0 [0.4 to 5.8] | 6.4 [3.1 to 11.4] | 5.1 [2.2 to 9.7]
  Redness: Moderate | 4.5 [1.8 to 9.1] | 3.3 [1.1 to 7.5] | 2.0 [0.4 to 5.7] | 1.3 [0.2 to 4.7] | 2.0 [0.4 to 5.8] | 5.1 [2.2 to 9.8] | 3.2 [1.0 to 7.2]
  Redness: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 1.3 [0.2 to 4.5] | 0.6 [0.0 to 3.5]
  Swelling: Mild | 3.2 [1.1 to 7.4] | 6.5 [3.2 to 11.7] | 5.3 [2.3 to 10.2] | 2.0 [0.4 to 5.7] | 4.0 [1.5 to 8.6] | 7.6 [4.0 to 13.0] | 2.5 [0.7 to 6.4]
  Swelling: Moderate | 1.9 [0.4 to 5.6] | 4.6 [1.9 to 9.2] | 4.0 [1.5 to 8.5] | 1.3 [0.2 to 4.7] | 2.0 [0.4 to 5.8] | 4.5 [1.8 to 9.0] | 4.4 [1.8 to 8.9]
  Swelling: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0.6 [0.0 to 3.5] | 0 [0.0 to 2.3]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, vomiting, diarrhea, chills, new/worsened muscle pain and joint pain. These were recorded by participants in an e-diary. Fever was defined as oral temperature greater than or equal to (>=) 38.0 degrees Celsius (deg C) and categorized as mild: >=38.0 to 38.4 deg C, moderate: >38.4 to 38.9 deg C and severe: >38.9 to 40.0 deg C. Vomiting was categorized as mild: 1-2 times in 24 hours (h); moderate: >2 times in 24h; severe: required intravenous (IV) hydration. Diarrhea was categorized as mild: 2-3 loose stools in 24h; moderate: 4-5 loose stools in 24h and severe: 6 or more loose stools in 24h. Headache, fatigue, chills, new/worsened muscle pain and joint pain were categorized as mild: didn't interfere with activity; moderate: some interference with activity and severe: prevented daily routine activity.
Time Frame: Day 1 to Day 7 after Vaccination on Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV
Number analyzed (Participants) | 154 | 153 | 150 | 152 | 149 | 157 | 158
Percentage of participants
  Fever: Mild | 3.2 [1.1 to 7.4] | 2.0 [0.4 to 5.6] | 1.3 [0.2 to 4.7] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 1.3 [0.2 to 4.5] | 2.5 [0.7 to 6.4]
  Fever: Moderate | 0.6 [0.0 to 3.6] | 1.3 [0.2 to 4.6] | 0 [0.0 to 2.4] | 1.3 [0.2 to 4.7] | 0 [0.0 to 2.4] | 0.6 [0.0 to 3.5] | 1.9 [0.4 to 5.4]
  Fever: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.3] | 0 [0.0 to 2.3]
  Fatigue: Mild | 21.4 [15.2 to 28.8] | 17.0 [11.4 to 23.9] | 18.0 [12.2 to 25.1] | 15.8 [10.4 to 22.6] | 17.4 [11.7 to 24.5] | 17.2 [11.6 to 24.0] | 20.9 [14.8 to 28.1]
  Fatigue: Moderate | 19.5 [13.5 to 26.6] | 19.0 [13.1 to 26.1] | 16.7 [11.1 to 23.6] | 7.9 [4.1 to 13.4] | 10.7 [6.3 to 16.9] | 20.4 [14.4 to 27.5] | 24.1 [17.6 to 31.5]
  Fatigue: Severe | 1.3 [0.2 to 4.6] | 1.3 [0.2 to 4.6] | 0.7 [0.0 to 3.7] | 0.7 [0.0 to 3.6] | 0.7 [0.0 to 3.7] | 1.3 [0.2 to 4.5] | 1.9 [0.4 to 5.4]
  Headache: Mild | 16.2 [10.8 to 23.0] | 19.0 [13.1 to 26.1] | 14.0 [8.9 to 20.6] | 15.8 [10.4 to 22.6] | 10.1 [5.7 to 16.1] | 15.3 [10.0 to 21.9] | 11.4 [6.9 to 17.4]
  Headache: Moderate | 5.2 [2.3 to 10.0] | 5.9 [2.7 to 10.9] | 8.7 [4.7 to 14.4] | 3.3 [1.1 to 7.5] | 2.7 [0.7 to 6.7] | 8.3 [4.5 to 13.7] | 7.0 [3.5 to 12.1]
  Headache: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0.6 [0.0 to 3.5] | 0.6 [0.0 to 3.5]
  Vomiting: Mild | 1.3 [0.2 to 4.6] | 0 [0.0 to 2.4] | 1.3 [0.2 to 4.7] | 2.6 [0.7 to 6.6] | 0.7 [0.0 to 3.7] | 0.6 [0.0 to 3.5] | 1.3 [0.2 to 4.5]
  Vomiting: Moderate | 0.6 [0.0 to 3.6] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.3] | 0 [0.0 to 2.3]
  Vomiting: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.3] | 0 [0.0 to 2.3]
  Diarrhea: Mild | 5.8 [2.7 to 10.8] | 3.3 [1.1 to 7.5] | 4.0 [1.5 to 8.5] | 7.2 [3.7 to 12.6] | 7.4 [3.7 to 12.8] | 4.5 [1.8 to 9.0] | 10.1 [5.9 to 15.9]
  Diarrhea: Moderate | 5.2 [2.3 to 10.0] | 0 [0.0 to 2.4] | 1.3 [0.2 to 4.7] | 2.6 [0.7 to 6.6] | 2.0 [0.4 to 5.8] | 0 [0.0 to 2.3] | 1.9 [0.4 to 5.4]
  Diarrhea: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0.7 [0.0 to 3.6] | 0 [0.0 to 2.4] | 0 [0.0 to 2.3] | 0.6 [0.0 to 3.5]
  Chills: Mild | 7.1 [3.6 to 12.4] | 5.9 [2.7 to 10.9] | 6.7 [3.2 to 11.9] | 2.0 [0.4 to 5.7] | 2.0 [0.4 to 5.8] | 4.5 [1.8 to 9.0] | 5.7 [2.6 to 10.5]
  Chills: Moderate | 3.2 [1.1 to 7.4] | 2.0 [0.4 to 5.6] | 2.7 [0.7 to 6.7] | 2.0 [0.4 to 5.7] | 0 [0.0 to 2.4] | 5.1 [2.2 to 9.8] | 5.1 [2.2 to 9.7]
  Chills: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0.6 [0.0 to 3.5] | 0 [0.0 to 2.3]
  New or worsened muscle pain: Mild | 7.8 [4.1 to 13.2] | 5.9 [2.7 to 10.9] | 6.0 [2.8 to 11.1] | 3.9 [1.5 to 8.4] | 6.0 [2.8 to 11.2] | 8.3 [4.5 to 13.7] | 7.0 [3.5 to 12.1]
  New or worsened muscle pain: Moderate | 5.2 [2.3 to 10.0] | 4.6 [1.9 to 9.2] | 4.7 [1.9 to 9.4] | 5.9 [2.7 to 10.9] | 4.7 [1.9 to 9.4] | 5.1 [2.2 to 9.8] | 7.6 [4.0 to 12.9]
  New or worsened muscle pain: Severe | 0 [0.0 to 2.4] | 0.7 [0.0 to 3.6] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0.6 [0.0 to 3.5] | 0 [0.0 to 2.3]
  New or worsened joint pain: Mild | 4.5 [1.8 to 9.1] | 4.6 [1.9 to 9.2] | 1.3 [0.2 to 4.7] | 2.0 [0.4 to 5.7] | 0.7 [0.0 to 3.7] | 4.5 [1.8 to 9.0] | 5.1 [2.2 to 9.7]
  New or worsened joint pain: Moderate | 3.9 [1.4 to 8.3] | 2.6 [0.7 to 6.6] | 7.3 [3.7 to 12.7] | 3.9 [1.5 to 8.4] | 3.4 [1.1 to 7.7] | 5.7 [2.7 to 10.6] | 3.8 [1.4 to 8.1]
  New or worsened joint pain: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.4] | 0 [0.0 to 2.3] | 0.6 [0.0 to 3.5]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention were included in evaluation of this outcome measure.
Time Frame: Within 1 Month after Vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV
Number analyzed (Participants) | 154 | 153 | 150 | 152 | 149 | 157 | 158
Percentage of participants | 9.1 [5.1 to 14.8] | 8.5 [4.6 to 14.1] | 8.0 [4.2 to 13.6] | 7.2 [3.7 to 12.6] | 8.1 [4.2 to 13.6] | 8.9 [5.0 to 14.5] | 8.9 [4.9 to 14.4]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Vaccination
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event were included in this outcome measure.
Time Frame: Within 6 Months after Vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV
Number analyzed (Participants) | 154 | 153 | 150 | 152 | 149 | 157 | 158
Percentage of participants | 0.6 [0.0 to 3.6] | 1.3 [0.2 to 4.6] | 2.7 [0.7 to 6.7] | 1.3 [0.2 to 4.7] | 1.3 [0.2 to 4.8] | 0.6 [0.0 to 3.5] | 1.9 [0.4 to 5.4]

5. Primary Outcome: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Neutralizing Titers (NTs) for Respiratory Syncytial Virus Subgroup A (RSV A) at 1 Month After Vaccination: Group 1 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV A were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV A, calculated as ratio of GMTs of Group 1 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: Evaluable immunogenicity population (EIP)= randomized participants who were eligible; received study intervention(s) to which they were randomized; 1-month post-vaccination blood collected within 27-42 days post vaccination; no protocol violations from randomization till 1-month postvaccination blood draw; had at least 1 valid, determinate assay result 1 month post vaccination. "Number of Participants Analyzed" = participants with valid and determinate assay results in EIP.
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 151 | 147
Titer | 18284 [15576.6 to 21462.6] | 18498 [15570.0 to 21975.9]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — Null hypothesis(H0) to assess noninferiority with respect to RSVpreF was evaluated by following hypothesis for both RSV A and B as measured by NT: H0: ln(μ1)- ln(μ4) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, ln(μ1), ln(μ4) are natural log of geometric mean of NT 1 month after vaccination for Group 1, 4, respectively; Geometric mean ratio = 0.99, 97.5% CI 2-sided [0.782 to 1.249] — GMRs and 2-sided confidence intervals (CIs) were calculated by exponentiating mean differences of logarithms of titers (Intervention Group [Group 1] minus Reference Group [Group 4]) and corresponding CIs (based on the Student t distribution)

6. Primary Outcome: GMT and GMR of NTs for Respiratory Syncytial Virus Subgroup B (RSV B) at 1 Month After Vaccination: Group 1 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV B were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV B, calculated as ratio of GMTs of Group 1 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: EIP= randomized participants who were eligible; received study intervention(s) to which they were randomized; 1-month post-vaccination blood collected within 27-42 days post vaccination; no protocol violations from randomization till 1-month postvaccination blood draw; had at least 1 valid, determinate assay result 1 month post vaccination. "Number of Participants Analyzed" = participants with valid and determinate assay results in EIP.
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 151 | 147
Titer | 15014 [12543.8 to 17971.8] | 16677 [13884.0 to 20031.4]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Geometric mean ratio = 0.90, 97.5% CI 2-sided [0.697 to 1.162] — GMRs and 2-sided CIs were calculated by exponentiating mean differences of the logarithms of titers (Intervention Group [Group 1] minus Reference Group [Group 4]) and corresponding CIs (based on the Student t distribution)

7. Primary Outcome: GMT and GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5 at 1 Month After Vaccination: Group 1 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 Omicron BA.4/BA.5 were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5, calculated as ratio of GMTs of Group 1 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 151 | 145
Titer | 3083 [2476.7 to 3838.1] | 3667 [2861.9 to 4697.5]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to BNT162b2 was evaluated by following hypothesis for both SARS-CoV-2 Omicron BA.4/BA.5 strain and reference strain as measured by NT: H0: ln(μ1)- ln(μ3) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, and ln(μ1) and ln(μ3) are natural log of geometric mean of NT 1 month after vaccination for Group 1, 3, respectively; Geometric mean ratio = 0.84, 97.5% CI 2-sided [0.605 to 1.168] — GMRs and 2-sided CIs were calculated by exponentiating mean differences of the logarithms of titers (Intervention Group [Group 1] minus Reference Group [Group 3]) and corresponding CIs (based on the Student t distribution)

8. Primary Outcome: GMT and GMR of NTs for SARS-CoV-2 Reference Strain at 1 Month After Vaccination: Group 1 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 reference strain were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 reference strain calculated as ratio of GMTs of Group 1 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 151 | 145
Titer | 9849 [8497.6 to 11416.5] | 12439 [10185.9 to 15190.1]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; Geometric mean ratio = 0.79, 97.5% CI 2-sided [0.618 to 1.014] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 1] minus Reference Group [Group 3]) and the corresponding CIs (based on the Student t distribution)

9. Primary Outcome: GMT and GMR of the Strain-Specific Hemagglutination Inhibition (HAI) Titers (H1N1 A/Victoria) of QIV at 1 Month After Vaccination: Group 1 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (H1N1 A/Victoria) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (H1N1 A/Victoria), calculated as ratio of GMTs of Group 1 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 149 | 143
Titer | 70 [56.8 to 87.3] | 67 [54.1 to 82.0]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to QIV was evaluated by following hypothesis for each of 4 strains included in QIV as measured by HAI titer: H0: ln(μ1)- ln(μ5) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, and ln(μ1) and ln(μ5) are natural log of the geometric mean of HAI titers 1 month after vaccination for Group 1,5, respectively; Geometric mean ratio = 1.06, 97.5% CI 2-sided [0.785 to 1.423] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 1] minus Reference Group [Group 5]) and the corresponding CIs (based on the Student t distribution)

10. Primary Outcome: GMT and GMR of the Strain-Specific HAI Titers (H3N2 A/Darwin) of QIV at 1 Month After Vaccination: Group 1 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (H3N2 A/Darwin) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (H3N2 A/Darwin), calculated as ratio of GMTs of Group 1 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 149 | 144
Titer | 138 [117.3 to 162.3] | 122 [105.7 to 141.4]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; Geometric mean ratio = 1.13, 97.5% CI 2-sided [0.909 to 1.402] — [estimate comment as in outcome 9, analysis 1]

11. Primary Outcome: GMT and GMR of the Strain-Specific HAI Titers (B/Austria) of QIV at 1 Month After Vaccination: Group 1 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (B/Austria) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (B/Austria), calculated as ratio of GMTs of Group 1 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 149 | 143
Titer | 71 [57.5 to 88.8] | 68 [54.3 to 84.8]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; Geometric mean ratio = 1.05, 97.5% CI 2-sided [0.773 to 1.434] — [estimate comment as in outcome 9, analysis 1]

12. Primary Outcome: GMT and GMR of the Strain-Specific HAI Titers (B/Phuket) of QIV at 1 Month After Vaccination: Group 1 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (B/Phuket) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (B/Phuket), calculated as ratio of GMTs of Group 1 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 148 | 141
Titer | 30 [23.6 to 37.2] | 27 [21.5 to 33.3]
Statistical Analysis 1: Comparison: Group 1: [RSVpreF + BNT162b2] + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; Geometric mean ratio = 1.11, 97.5% CI 2-sided [0.807 to 1.515] — [estimate comment as in outcome 9, analysis 1]

13. Primary Outcome: GMT and GMR of NTs for RSV A at 1 Month After Vaccination: Group 2 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV A were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV A, calculated as ratio of GMTs of Group 2 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: EIP= randomized participants who were eligible; received study intervention(s) to which they were randomized; 1-month post-vaccination blood collected within 27-42 days post vaccination; no protocol violations from randomization till 1-month postvaccination blood draw; had at least 1 valid, determinate assay result 1 month post vaccination.
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 148 | 147
Titer | 18414 [15172.8 to 22346.9] | 18498 [15570.0 to 21975.9]
Statistical Analysis 1: Comparison: Group 2: [RSVpreF+BNT162b2] + Placebo vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — Null hypothesis(H0) to assess noninferiority with respect to RSVpreF was evaluated by following hypothesis for both RSV A, RSV B as measured by NT:H0: ln(μ2)- ln(μ4) <=ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority and ln(μ2) and ln(μ4) are natural log of geometric mean of NT 1 month after vaccination for Group 2, 4, respectively; Geometric mean ratio = 1.00, 97.5% CI 2-sided [0.769 to 1.288] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 2] minus Reference Group [Group 4]) and the corresponding CIs (based on the Student t distribution)

14. Primary Outcome: GMT and GMR of NTs for RSV B at 1 Month After Vaccination: Group 2 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV B were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV B, calculated as ratio of GMTs of Group 2 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 13
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 148 | 147
Titer | 18227 [14961.9 to 22204.2] | 16677 [13884.0 to 20031.4]
Statistical Analysis 1: Comparison: Group 2: [RSVpreF+BNT162b2] + Placebo vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Geometric mean ratio = 1.09, 97.5% CI 2-sided [0.836 to 1.429] — [estimate comment as in outcome 13, analysis 1]

15. Primary Outcome: GMT and GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5 at 1 Month After Vaccination: Group 2 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 Omicron BA.4/BA.5 were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5, calculated as ratio of GMTs of Group 2 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 147 | 145
Titer | 3083 [2412.5 to 3940.4] | 3667 [2861.9 to 4697.5]
Statistical Analysis 1: Comparison: Group 2: [RSVpreF+BNT162b2] + Placebo vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to BNT162b2 will be evaluated by following hypothesis for both SARS-CoV-2 Omicron BA.4/BA.5 strain and reference strain as measured by NT:H0: ln(μ2)- ln(μ3) <= ln(0.5)where ln(0.5) corresponds to a 2-fold margin for noninferiority and ln(μ2) and ln(μ3) are natural log of geometric mean of NT 1 month after vaccination for Group 2,3, respectively; Geometric mean ratio = 0.84, 97.5% CI 2-sided [0.594 to 1.190] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 2] minus Reference Group [Group 3]) and the corresponding CIs (based on the Student t distribution)

16. Primary Outcome: GMT and GMR of NTs for SARS-CoV-2 Reference Strain at 1 Month After Vaccination: Group 2 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 reference strain were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 reference strain calculated as ratio of GMTs of Group 2 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 13
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 148 | 145
Titer | 10489 [8500.2 to 12943.5] | 12439 [10185.9 to 15190.1]
Statistical Analysis 1: Comparison: Group 2: [RSVpreF+BNT162b2] + Placebo vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Geometric mean ratio = 0.84, 97.5% CI 2-sided [0.632 to 1.125] — [estimate comment as in outcome 15, analysis 1]

17. Secondary Outcome: GMT and GMR of NTs for RSV A at 1 Month After Vaccination: Group 7 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV A were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV A, calculated as ratio of GMTs of Group 7 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 13
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 154 | 147
Titer | 26303 [22338.8 to 30970.5] | 18498 [15570.0 to 21975.9]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — Null hypothesis(H0) to assess noninferiority with respect to RSVpreF was evaluated by following hypothesis for both RSV A and B as measured by NT: H0: ln(μ1)- ln(μ4) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, ln(μ1), ln(μ4) are natural log of geometric mean of NT 1 month after vaccination for Group 7, 4, respectively; Geometric mean ratio = 1.42, 97.5% CI 2-sided [1.123 to 1.801] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 7] minus Reference Group [Group 4]) and the corresponding CIs (based on the Student t distribution)

18. Secondary Outcome: GMT and GMR of NTs for RSV B at 1 Month After Vaccination: Group 7 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV B were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV B, calculated as ratio of GMTs of Group 7 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 13
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 154 | 147
Titer | 21182 [17525.4 to 25600.8] | 16677 [13884.0 to 20031.4]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — [test comment as in outcome 17, analysis 1]; Geometric mean ratio = 1.27, 97.5% CI 2-sided [0.977 to 1.651] — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: GMT and GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5 at 1 Month After Vaccination: Group 7 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 Omicron BA.4/BA.5 were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5, calculated as ratio of GMTs of Group 7 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 153 | 145
Titer | 3148 [2482.6 to 3992.0] | 3667 [2861.9 to 4697.5]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to BNT162b2 will be evaluated by following hypothesis for both SARS-CoV-2 Omicron BA.4/BA.5 strain and reference strain as measured by NT:H0: ln(μ2)- ln(μ3) <= ln(0.5)where ln(0.5) corresponds to a 2-fold margin for noninferiority and ln(μ2) and ln(μ3) are natural log of geometric mean of NT 1 month after vaccination for Group 7,3, respectively; Geometric mean ratio = 0.86, 97.5% CI 2-sided [0.610 to 1.208] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 7] minus Reference Group [Group 3]) and the corresponding CIs (based on the Student t distribution)

20. Secondary Outcome: GMT and GMR of NTs for SARS-CoV-2 Reference Strain at 1 Month After Vaccination: Group 7 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 reference strain were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 reference strain calculated as ratio of GMTs of Group 7 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 153 | 145
Titer | 12588 [10312.2 to 15365.4] | 12439 [10185.9 to 15190.1]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to BNT162b2 was evaluated by following hypothesis for both SARS-CoV-2 Omicron BA.4/BA.5 strain and reference strain as measured by NT: H0: ln(μ1)- ln(μ3) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, and ln(μ1) and ln(μ3) are natural log of geometric mean of NT 1 month after vaccination for Group 7, 3, respectively; Geometric mean ratio = 1.01, 97.5% CI 2-sided [0.764 to 1.340] — [estimate comment as in outcome 19, analysis 1]

21. Secondary Outcome: GMT and GMR of the Strain-Specific HAI Titers (H1N1 A/Victoria) of QIV at 1 Month After Vaccination: Group 7 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (H1N1 A/Victoria) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (H1N1 A/Victoria), calculated as ratio of GMTs of Group 7 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 152 | 143
Titer | 166 [141.0 to 194.7] | 67 [54.1 to 82.0]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to QIV was evaluated by following hypothesis for each of 4 strains included in QIV as measured by HAI titer: H0: ln(μ1)- ln(μ5) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, and ln(μ1) and ln(μ5) are natural log of the geometric mean of HAI titers 1 month after vaccination for Group 7,5, respectively; Geometric mean ratio = 2.49, 97.5% CI 2-sided [1.914 to 3.232] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 7] minus Reference Group [Group 5]) and the corresponding CIs (based on the Student t distribution)

22. Secondary Outcome: GMT and GMR of the Strain-Specific HAI Titers (H3N2 A/Darwin) of QIV at 1 Month After Vaccination: Group 7 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (H3N2 A/Darwin) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (H3N2 A/Darwin), calculated as ratio of GMTs of Group 7 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 151 | 144
Titer | 159 [135.6 to 186.5] | 122 [105.7 to 141.4]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 1]; Geometric mean ratio = 1.30, 97.5% CI 2-sided [1.049 to 1.612] — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: GMT and GMR of the Strain-Specific HAI Titers (B/Austria) of QIV at 1 Month After Vaccination: Group 7 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (B/Austria) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (B/Austria), calculated as ratio of GMTs of Group 7 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 150 | 143
Titer | 107 [85.8 to 134.4] | 68 [54.3 to 84.8]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 1]; Geometric mean ratio = 1.58, 97.5% CI 2-sided [1.155 to 2.165] — [estimate comment as in outcome 21, analysis 1]

24. Secondary Outcome: GMT and GMR of the Strain-Specific HAI Titers (B/Phuket) of QIV at 1 Month After Vaccination: Group 7 Versus Group 5
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for hemagglutination inhibition titers (B/Phuket) were reported in the descriptive data section of this outcome measure. GMR of NTs for hemagglutination inhibition titers (B/Phuket), calculated as ratio of GMTs of Group 7 to Group 5, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 7: RSVpreF + BNT162b2 + QIV | Group 5: QIV + Placebo
Number analyzed (Participants) | 149 | 141
Titer | 93 [78.5 to 111.0] | 27 [21.5 to 33.3]
Statistical Analysis 1: Comparison: Group 7: RSVpreF + BNT162b2 + QIV vs Group 5: QIV + Placebo; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 1]; Geometric mean ratio = 3.49, 97.5% CI 2-sided [2.640 to 4.604] — [estimate comment as in outcome 21, analysis 1]

25. Secondary Outcome: GMT and GMR of NTs for RSV A at 1 Month After Vaccination: Group 6 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV A were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV A, calculated as ratio of GMTs of Group 6 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 6: RSVpreF + BNT162b2 + Placebo | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 149 | 147
Titer | 26452 [22515.2 to 31076.8] | 18498 [15570.0 to 21975.9]
Statistical Analysis 1: Comparison: Group 6: RSVpreF + BNT162b2 + Placebo vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — Null hypothesis(H0) to assess noninferiority with respect to RSVpreF was evaluated by following hypothesis for both RSV A and B as measured by NT: H0: ln(μ1)- ln(μ4) <= ln(0.5) where ln(0.5) corresponds to a 2-fold margin for noninferiority, ln(μ1), ln(μ4) are natural log of geometric mean of NT 1 month after vaccination for Group 6, 4, respectively; Geometric mean ratio = 1.43, 97.5% CI 2-sided [1.131 to 1.808] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 6] minus Reference Group [Group 4]) and the corresponding CIs (based on the Student t distribution)

26. Secondary Outcome: GMT and GMR of NTs for RSV B at 1 Month After Vaccination: Group 6 Versus Group 4
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for RSV B were reported in the descriptive data section of this outcome measure. GMR of NTs for RSV B, calculated as ratio of GMTs of Group 6 to Group 4, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 6: RSVpreF + BNT162b2 + Placebo | Group 4: RSVpreF + Placebo
Number analyzed (Participants) | 148 | 147
Titer | 22859 [19040.4 to 27442.5] | 16677 [13884.0 to 20031.4]
Statistical Analysis 1: Comparison: Group 6: RSVpreF + BNT162b2 + Placebo vs Group 4: RSVpreF + Placebo; Test type: Non-Inferiority — [test comment as in outcome 25, analysis 1]; Geometric mean ratio = 1.37, 97.5% CI 2-sided [1.060 to 1.773] — [estimate comment as in outcome 25, analysis 1]

27. Secondary Outcome: GMT and GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5 at 1 Month After Vaccination: Group 6 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 Omicron BA.4/BA.5 were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 Omicron BA.4/BA.5, calculated as ratio of GMTs of Group 6 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 6: RSVpreF + BNT162b2 + Placebo | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 148 | 145
Titer | 3430 [2756.9 to 4267.7] | 3667 [2861.9 to 4697.5]
Statistical Analysis 1: Comparison: Group 6: RSVpreF + BNT162b2 + Placebo vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — Null hypothesis (H0) to assess noninferiority with respect to BNT162b2 will be evaluated by following hypothesis for both SARS-CoV-2 Omicron BA.4/BA.5 strain and reference strain as measured by NT:H0: ln(μ2)- ln(μ3) <= ln(0.5)where ln(0.5) corresponds to a 2-fold margin for noninferiority and ln(μ2) and ln(μ3) are natural log of geometric mean of NT 1 month after vaccination for Group 6,3, respectively; Geometric mean ratio = 0.94, 97.5% CI 2-sided [0.673 to 1.300] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences of the logarithms of the titers (Intervention Group [Group 6] minus Reference Group [Group 3]) and the corresponding CIs (based on the Student t distribution)

28. Secondary Outcome: GMT and GMR of NTs for SARS-CoV-2 Reference Strain at 1 Month After Vaccination: Group 6 Versus Group 3
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). GMTs of NTs for SARS-CoV-2 reference strain were reported in the descriptive data section of this outcome measure. GMR of NTs for SARS-CoV-2 reference strain calculated as ratio of GMTs of Group 6 to Group 3, was reported in the statistical analysis section.
Time Frame: 1 Month after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titer
Arm/Group | Group 6: RSVpreF + BNT162b2 + Placebo | Group 3: BNT162b2 + Placebo
Number analyzed (Participants) | 148 | 145
Titer | 12111 [10010.3 to 14652.1] | 12439 [10185.9 to 15190.1]
Statistical Analysis 1: Comparison: Group 6: RSVpreF + BNT162b2 + Placebo vs Group 3: BNT162b2 + Placebo; Test type: Non-Inferiority — [test comment as in outcome 27, analysis 1]; Geometric mean ratio = 0.97, 97.5% CI 2-sided [0.740 to 1.281] — [estimate comment as in outcome 27, analysis 1]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: From Day 1 to Day 7 after Vaccination 1; Non serious AEs: up to 1 month after Vaccination 1, SAEs: up to 6 months after Vaccination 1
Description: Same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included all participants who received the study intervention.
Arm/Group | Group 1: [RSVpreF + BNT162b2] + QIV | Group 2: [RSVpreF+BNT162b2] + Placebo | Group 3: BNT162b2 + Placebo | Group 4: RSVpreF + Placebo | Group 5: QIV + Placebo | Group 6: RSVpreF + BNT162b2 + Placebo | Group 7: RSVpreF + BNT162b2 + QIV
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/153 | 0/150 | 0/152 | 0/149 | 0/157 | 0/158
Serious Adverse Events (participants affected / at risk) | 1/154 | 2/153 | 4/150 | 2/152 | 2/149 | 1/157 | 3/158
Other Adverse Events (participants affected / at risk) | 114/154 | 107/153 | 110/150 | 73/152 | 96/149 | 114/157 | 122/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: [RSVpreF + BNT162b2] + QIV (N=154) | Group 2: [RSVpreF+BNT162b2] + Placebo (N=153) | Group 3: BNT162b2 + Placebo (N=150) | Group 4: RSVpreF + Placebo (N=152) | Group 5: QIV + Placebo (N=149) | Group 6: RSVpreF + BNT162b2 + Placebo (N=157) | Group 7: RSVpreF + BNT162b2 + QIV (N=158)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebellar ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle cerebral artery stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thalamic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: [RSVpreF + BNT162b2] + QIV (N=154) | Group 2: [RSVpreF+BNT162b2] + Placebo (N=153) | Group 3: BNT162b2 + Placebo (N=150) | Group 4: RSVpreF + Placebo (N=152) | Group 5: QIV + Placebo (N=149) | Group 6: RSVpreF + BNT162b2 + Placebo (N=157) | Group 7: RSVpreF + BNT162b2 + QIV (N=158)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 17 | 5 | 8 | 16 | 14 | 7 | 20
Vomiting (VOMITING) (Gastrointestinal disorders) | 3 | 0 | 2 | 4 | 1 | 1 | 2
Chills (CHILLS) (General disorders) | 16 | 12 | 14 | 6 | 3 | 16 | 17
Fatigue (FATIGUE) (General disorders) | 65 | 57 | 53 | 37 | 43 | 61 | 74
Injection site erythema (REDNESS) (General disorders) | 12 | 14 | 11 | 4 | 6 | 20 | 14
Injection site pain (PAIN AT THE INJECTION SITE) (General disorders) | 88 | 80 | 94 | 16 | 77 | 89 | 85
Injection site swelling (SWELLING) (General disorders) | 8 | 17 | 14 | 5 | 9 | 20 | 11
Pyrexia (FEVER) (General disorders) | 6 | 5 | 2 | 2 | 0 | 3 | 7
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 3 | 1
Arthralgia (NEW OR WORSENED JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 13 | 11 | 13 | 9 | 6 | 16 | 15
Myalgia (NEW OR WORSENED MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 20 | 17 | 16 | 15 | 16 | 22 | 23
Headache (HEADACHE) (Nervous system disorders) | 33 | 38 | 34 | 29 | 19 | 38 | 30
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT05886777/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05886777/SAP_001.pdf